CLINICAL TRIAL: NCT04930887
Title: Prospective, Randomized, Double-blinded, Placebo-controlled, Cross-over Trial of Endoscopically Guided Injection of Exparel (Bupivacaine) Towards the Ipsilateral Pterygopalatine Fossa for the Treatment of Craniofacial Pain
Brief Title: Clinical Trial of Endoscopically Guided Injection of Exparel (Bupivacaine) for the Treatment of Craniofacial Pain
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Peter Hwang, PROFESSOR OF OTOLARYNGOLOGY - HEAD & NECK SURGERY (OHNS) AND, BY COURTESY, OF NEUROSURGERY AT THE STANFORD UNIVERSITY MEDICAL CENTER, Stanford University
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 60832
Record Dates: First submitted 2021-06-11; First posted 2021-06-18 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Craniofacial Pain; Migraine; Cluster Headache; Trigeminal Autonomic Cephalgia; Sphenopalatine Ganglion Neuralgia; Paroxysmal Hemicrania
MeSH Terms: conditions — Facial Pain; Migraine Disorders; Cluster Headache; Trigeminal Autonomic Cephalalgias; Facial Neuralgia; Paroxysmal Hemicrania | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Exparel (Active Comparator): Patients receive an endoscopically guided injection of Exparel (Bupivacaine).
  Interventions: Drug: Exparel (Bupivacaine Liposome)
- Saline (Placebo Comparator): Patients receive an endoscopically guided injection of saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: Exparel (Bupivacaine Liposome) — Non-opioid postsurgical analgesic used in the management of postsurgical pain; 133 mg/10 mL (13.3 mg/mL) single-dose vial (per Pacira), study administers 3cc bilaterally
  Arms: Exparel
Drug: Saline — Prescription medicine used for fluid and electrolyte replenishment for intravenous administration; Exparel-matched Placebo treatment
  Arms: Saline

SUMMARY:
Exparel has a proven efficacy in providing pain relief for up to 72 hours with a single-dose administration at surgical sites. The study aims to evaluate the effectiveness of endoscopically-guided injection of Exparel (Bupivacaine) for the treatment of craniofacial pain. This study would be conducted in a prospective, randomized, double-blinded, placebo- controlled, and cross-over fashion. We aim to investigate whether the administration of Exparel (Bupivacaine) to the lateral nasal wall may positively impact craniofacial pain and functional outcomes, in patients who experience relief with the topical application of Lidocaine (routinely given prior to almost all ENT endoscopy).

ELIGIBILITY:
Inclusion Criteria:

* Patients with a chief complaint of craniofacial pain (migraine, cluster headache, trigeminal autonomic cephalgia, sphenopalatine ganglioneuraligia, paroxysmal hemicrania) who has Stanford Pain & ENT clinic visit

Exclusion Criteria:

* age <18 or >80
* pregnant women
* economically disadvantaged (not able to afford clinic visits/treatments)
* decisionally impaired (unable to obtain informed consent)
* has allergy to bupivacaine
* unable or unwilling to participate plans to participate in another clinical study at any time during this study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-02-01 (Actual); Primary Completion 2025-06 (Estimated); Study Completion 2030-06 (Estimated)

PRIMARY OUTCOMES:
Change of Pain Score | Baseline to day 21
  Scores range from 0-10 (0=no pain, 10=worst pain)

SECONDARY OUTCOMES:
Change of Associated Symptoms | Baseline to day 21
  Changes of associated symptoms, including nausea, photophobia, use of rescue medication, relapse of headache, and/or change in headache disability scores

CONTACTS AND LOCATIONS:
Overall Officials: Peter Hwang, MD, Principal Investigator — Stanford University
Locations (1):
- Peter H Hwang, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No
IPD will be kept confidential and private and won't be used for any other studies or shared with other researchers.